CLINICAL TRIAL: NCT01132729
Title: A Single Dose, 2-Period, 2-Treatment 2-Way Crossover Bioequivalency Study of Valacyclovir Caplets Under Fasting Conditions
Brief Title: Bioequivalency Study of Valacyclovir Hydrochloride 1000 mg Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: VALA-T1000-PVFS-1
Record Dates: First submitted 2010-05-25; First posted 2010-05-28 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Herpes Zoster; Shingles; Genital Herpes
MeSH Terms: conditions — Herpes Zoster; Herpes Genitalis | interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Valacyclovir Hydrochloride — 1000 mg caplet
  Other Names: Valtrex

SUMMARY:
The objective of this study was to prove the bioequivalence of Valacyclovir Hydrochlorothiazide Caplet under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to valacyclovir hydrochloride or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2006-09; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Alan Copa, PharmD, Principal Investigator — PRACs Institute, Ltd.
Locations (1):
- PRACs Institute, Ltd., Fargo, North Dakota, United States